CLINICAL TRIAL: NCT04978714
Title: Prevalence of Urodynamic Stress Incontinence and/or Detrusor Overactivity in Women With Cystocele and the Changes of Continence Function After Cystocele Repair
Brief Title: USI and/or DO in Women With Cystocele Before and After Cystocele Repair
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202105056RINC
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Urodynamic Stress Incontinence; Detrusor Overactivity
Keywords: Urodynamic stress incontinence; Detrusor Overactivity; Cystocele
MeSH Terms: conditions — Urinary Bladder, Overactive; Cystocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with cystocele: All women with ≥ stage II cystocele who visited the urogynecological department of a medical center for cystocele repair
  Interventions: Procedure: Cystocele repair

INTERVENTIONS:
Procedure: Cystocele repair — Fascial repair for endopelvic fascia and anterior colporrhaphy

SUMMARY:
The changes of lower urinary tract function after cystocele repair are important for perioperative consultation and management. Thus, the aim of this retrospective study was to evaluate the prevalence of urodynamic stress incontinence and/or detrusor overactivity in women with ≥ stage II cystocele and the changes of incontinence function after cystocele repair.

DETAILED DESCRIPTION:
Between November 2010 and October 2020, all women with ≥ stage II cystocele who visited the urogynecological department of a medical center for cystocele repair were reviewed. Those women who had complete data of preoperative and postoperative 3-month follow-up urodynamic data were excluded from this study. Urodynamic stress incontinence was diagnosed by the finding of involuntary leakage during filling cystometry or stress urethral pressure profile, associated with increased intra-abdominal pressure, in the absence of a detrusor contraction. Detrusor overactivity was defined as the occurrence of involuntary detrusor contractions during filling cytometry.

STATA software was used for statistical analysis. Chi2 test, univariate and multivariable logistic regression tests were used for statistical analysis as appropriate. A p < 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with ≥ stage II cystocele
* Received cystocele repair
* Complete urodynamic study before and after surgery

Exclusion Criteria:

* Incomplete data
* Chronic infection
* Recurrent surgery for cystocele

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with ≥ stage II cystocele who visited the urogynecological department of a medical center for cystocele repair
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Urodynamic stress incontinence | November 2010 and October 2020
  the finding of involuntary leakage during filling cystometry or stress urethral pressure profile, associated with increased intra-abdominal pressure, in the absence of a detrusor contraction
Detrusor overactivity | November 2010 and October 2020
  the occurrence of involuntary detrusor contractions during filling cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data is available under reasonable request

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Lamblin G, Delorme E, Cosson M, Rubod C. Cystocele and functional anatomy of the pelvic floor: review and update of the various theories. Int Urogynecol J. 2016 Sep;27(9):1297-305. doi: 10.1007/s00192-015-2832-4. Epub 2015 Sep 4. PMID 26337427
- [Result] Leron E, Weintraub AY, Mastrolia SA, Schwarzman P. Overactive Bladder Syndrome: Evaluation and Management. Curr Urol. 2018 Mar;11(3):117-125. doi: 10.1159/000447205. Epub 2018 Feb 20. PMID 29692690
- [Result] Hsiao SM, Lin HH, Kuo HC. Videourodynamic Studies of Women with Voiding Dysfunction. Sci Rep. 2017 Jul 28;7(1):6845. doi: 10.1038/s41598-017-07163-2. PMID 28754926
- [Result] Hsiao SM, Chang TC, Wu PC, Lin HH. Predictors of an improvement in the severity of concomitant urodynamic stress incontinence after transvaginal mesh surgery for pelvic organ prolapse. J Formos Med Assoc. 2020 May;119(5):917-924. doi: 10.1016/j.jfma.2019.12.016. Epub 2020 Mar 5. PMID 32146026
- [Result] Huang WC, Yang SH, Yang JM. Clinical Importance and Surgical Outcomes of Green Type III Cystocele in Women With Anterior Vaginal Prolapse. J Ultrasound Med. 2015 Dec;34(12):2279-85. doi: 10.7863/ultra.14.11066. Epub 2015 Nov 16. PMID 26573101